CLINICAL TRIAL: NCT05554185
Title: Effects of Probiotic Supplementation During Pregnancy on Maternal and Infant Outcomes in Preeclampsia High-risk Groups Based on Abnormal Intestinal Flora: a Randomized Controlled Clinical Trial
Brief Title: Probiotic Supplementation During Pregnancy in Preeclampsia High-risk Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NFEC-2022-358
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: PE (Pre-eclampsia) High-risk Population With Gut Microbiota Dysbiosis During Their Pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): aspirin 100mg and probiotics 1 bag
  Interventions: Dietary Supplement: aspirin 100mg and probiotics 1 bag
- group B (Placebo Comparator): aspirin 100mg and placebo1 bag
  Interventions: Dietary Supplement: aspirin 100mg and probiotics 1 bag

INTERVENTIONS:
Dietary Supplement: aspirin 100mg and probiotics 1 bag — taking aspirin 100mg and probiotics 1 bag per day from 14-16 weeks of pregnancy until 35 + 6 weeks of pregnancy or emergency delivery.

SUMMARY:
In this randomized controlled study, preventive intervention of aspirin combined with probiotics or aspirin combined with placebo would given to PE (pre-eclampsia) high-risk population with gut microbiota dysbiosis during their pregnancy, and finally assess the efficacy and safety of aspirin combined with probiotics to prevent PE.

ELIGIBILITY:
Inclusion Criteria:

* PE high-risk population aged 18-50 years with gut microbiota dysbiosis
* No severe cardiopulmonary diseases
* No severe hepatic and renal insufficiency
* No severe active infection
* Pregnant women did not take antibiotics or antifungal drugs 30 days before fecal sample collection; No probiotic preparation was taken 2 weeks before sample collection; Never take drugs that may interfere with glucose and lipid metabolism
* No diseases affecting intestinal microecology
* No history of smoking and drinking
* The researchers evaluated those pregnant women expected to deliver more than 20 weeks
* Voluntarily participate in this clinical study and sign the informed consent form

Exclusion Criteria:

* With severe cardiopulmonary, hepatic and renal insufficiency
* With uncontrolled active infections 2 weeks before enrollment
* Subjects took antibiotics or antifungal drugs 30 days before sample collection; Take probiotics 2 weeks before sample collection; Have taken drugs that may interfere with glucose and lipid metabolism
* with diseases affecting intestinal microecology
* Smoking and drinking history
* With acute gastrointestinal ulcer
* Hemorrhagic constitution
* Other discomfort assessed by the investigato

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 338 (Estimated)
Dates: Start 2022-09-21 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of preeclampsia | From being recruited to 6 weeks after delivery
  After 20 weeks of pregnancy, systolic blood pressure ≥ 140mmHg and / or diastolic blood pressure ≥ 90mmHg, accompanied by any of the following items: urinary protein ≥ 0.3g/24h, or urinary protein / creatinine ratio ≥ 0.3,or random urinary protein ≥ (+) (examination method for unconditional protein quantification); Non-albuminuria can be accompanied by any kind of organ or system involvement: heart, lung, liver, kidney and other important organs, or abnormal changes in blood system, digestive system, nervous system, placenta-fetus, etc.

SECONDARY OUTCOMES:
The incidence of fetal growth restriction | From being recruited to 6 weeks after delivery
  due to the influence of pathological factors such as mother, fetus and placenta, fetal growth does not reach its due genetic potential, which is characterized by fetal body weight or abdominal circumference estimated by ultrasound lower than the 10th percentile of the corresponding gestational age

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen X, Li P, Liu M, Zheng H, He Y, Chen MX, Tang W, Yue X, Huang Y, Zhuang L, Wang Z, Zhong M, Ke G, Hu H, Feng Y, Chen Y, Yu Y, Zhou H, Huang L. Gut dysbiosis induces the development of pre-eclampsia through bacterial translocation. Gut. 2020 Mar;69(3):513-522. doi: 10.1136/gutjnl-2019-319101. Epub 2020 Jan 3. PMID 31900289